CLINICAL TRIAL: NCT06539767
Title: Risk Assessment and Mechanism Analysis of Intracranial Multiple Aneurysm Instability Based on High-resolution Magnetic Resonance, Imaging Histology and Hemodynamics
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-KY-127-01
Record Dates: First submitted 2024-06-04; First posted 2024-08-06 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Arterial Aneurysm Wall Enhancement on HRMRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project proposes to establish a prospective cohort of MIA based on a preexisting multicenter MIA database and to combine multidimensional methods such as high-resolution magnetic resonance, hemodynamics, ambulatory blood pressure, and imaging histology to study aneurysm instability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, male or infertile female;
* Diagnosed as IA (intracranial aneurysm) through CTA, MRA, or DSA; And it is suitable for endovascular intervention treatment
* The patient and/or their legal representative or guardian fully understand the research purpose, voluntarily participate and sign informed consent Books;
* Patients willing to cooperate with high-resolution magnetic resonance imaging.
* Patients willing to follow up and evaluate according to clinical research protocol requirements

Exclusion Criteria:

* AVM (arteriovenous malformation), Moyamoya disease, or DAVF (dural arteriovenous fistula) related aneurysms;
* Patients with contraindications for high-resolution magnetic resonance imaging;
* Participants in clinical trials of other drugs or medical devices;
* Patients with severe underlying diseases and extremely poor clinical conditions who cannot tolerate general anesthesia surgery;
* Patients with poor compliance and inability to cooperate with follow-up;
* Possible or clear history of severe allergy to contrast agents;
* Patients with a life expectancy of less than 2 years;
* Women who are breastfeeding and preparing for pregnancy during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  1. be older than 18 years of age; 2. complete a high-resolution magnetic resonance exam
  Exclusion Criteria:
  1. aneurysm combined with other cerebrovascular diseases; 2. substandard image quality
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
High resolution MRI aneurysm features | 1 year
  Enhancement grade was defined as follows: grade 0 for none enhancement, grade 1 for focal enhancement, involved the neck, the intermediate portion, the dome, or a bleb;grade 2 for thin annular enhancement (maximum thickness≤1 mm) , grade 3 for thick annular enhancement(maximum thickness>1 mm) .

SECONDARY OUTCOMES:
postoperative mRS score | 1 year
  MRS score definition: The MRS score, also known as the Modified Rankin Scale, is a scale used to evaluate the neurological recovery status of stroke patients. It is divided into seven levels, Level 0: completely asymptomatic. Level 1: Despite symptoms, without obvious disabilities, able to complete all frequently engaged work and activities.
  Level 2: Mild disability, unable to complete all work and activities, but able to handle personal affairs without the need for assistance from others.
  Level 3: Moderate disability, requiring assistance from others to walking without assistance.
  Level 4: Severe disability, unable to walk without the help of others, unable to take care of one's own needs.
  Level 5: Severe disability, bedridden, urinary and fecal incontinence, requiring continuous care, and requiring multiple 24-hour care from others.
  Level 6: Death. The higher the mRS score, the worse the patient's prognosis.
postoperative aneurysm occlusion rate | 1 year
  Raymond classification, grade I: complete embolism; Grade II: residual aneurysm neck;

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhujiang Hospital, Guangzhou, Guangdong
  - Southern medical university, zhujiang hospital, Guangzhou